CLINICAL TRIAL: NCT04721509
Title: Effect of Smartphone Based Telemedicine and Education in Patients With Type 1 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 4-2020-0880
Record Dates: First submitted 2021-01-21; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes Mellitus, Telemedicine, Smartphone, Type 1, Child, Adolescent, Young Adult
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Inclusion criteria: patients with type 1 diabetes with A1c>8.0% Exclusion criteria: chronic disease, psychological disease, children aged under 12 with parents with psychological disease, athletics Method: We divide subjects as an experimental group and a control group by randomization, and they visit outpatient clinic every 12 weeks. We perform telemedicine and education with smartphone application to the experimental group every 2 weeks. We evaluate the effect of smartphone based telemedicine and education in patients with type 1 diabetes mellitus with checking A1c and checklist at baseline, 12 weeks and 24 weeks after starting of the research.
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone-based telemedicine (Experimental)
  Interventions: Device: Experimental : Smartphone-based telemedicine with the app 'Songaree diabetes'
- Conventional management without telemedicine (No Intervention)

INTERVENTIONS:
Device: Experimental : Smartphone-based telemedicine with the app 'Songaree diabetes' — Experimental group: outpatient clinic and offline education every 12 weeks plus telemedicine and education with smartphone app 'Songaree diabetes' every 2 weeks for 24 weeks
  Arms: Smartphone-based telemedicine

SUMMARY:
Objective: evaluation of effect of smartphone based telemedicine and education in patients with type 1 diabetes mellitus Outline: Among the patients with type 1 diabetes, the group with telemedicine and education using smartphone set as a experimental group and the group without those set as a control group, respectively.

Sample size: experimental group (n=50), control group (n=50) Inclusion criteria: patients with type 1 diabetes with A1c>8.0% Exclusion criteria: chronic disease, psychological disease, children aged under 12 with parents with psychological disease, athletics Method: We divide subjects as an experimental group and a control group by randomization, and they visit outpatient clinic every 12 weeks. We perform telemedicine and education with smartphone application to the experimental group every 2 weeks. We evaluate the effect of smartphone based telemedicine and education in patients with type 1 diabetes mellitus with checking A1c and checklist at baseline, 12 weeks and 24 weeks after starting of the research.

Variables: A1c, satisfaction, knowledge, self-confidence, willing to continuing, quality of life, physical activity, drinking, smoking Primary endpoint: Improvement in HbA1c of experimental group Secondary endpoint: No improvement in HbA1c of control group

ELIGIBILITY:
Inclusion Criteria:

a. patients aged under 30 with type 1 diabetes b. patients who control glucose level with multiple daily injection of insulin pump c. Patients who agree the task to check glucose level during the experiment d. patients who has been diagnosed as type 1 diabetes more than 3 months e. patients whose A1c more than 8.0% within 6 months f. Patients who can use smartphone all day 2) exclusion criteria

1. chronic disease (except thyroid disorders with euthyroidism), psychological disease
2. Patients aged under 12 whose parents have psychological disease
3. Patients who cannot use smartphone app properly
4. athletics
5. Patients who use continuous glucose monitoring

Exclusion Criteria:

-

Ages: 0 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
change in HbA1c of experimental group | 6 months

SECONDARY OUTCOMES:
No change in HbA1c of control group | 6 months later

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Seong Kim, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maahs DM, West NA, Lawrence JM, Mayer-Davis EJ. Epidemiology of type 1 diabetes. Endocrinol Metab Clin North Am. 2010 Sep;39(3):481-97. doi: 10.1016/j.ecl.2010.05.011. PMID 20723815
- [Result] Song SO, Song YD, Nam JY, Park KH, Yoon JH, Son KM, Ko Y, Lim DH. Epidemiology of Type 1 Diabetes Mellitus in Korea through an Investigation of the National Registration Project of Type 1 Diabetes for the Reimbursement of Glucometer Strips with Additional Analyses Using Claims Data. Diabetes Metab J. 2016 Feb;40(1):35-45. doi: 10.4093/dmj.2016.40.1.35. PMID 26912154
- [Result] American Diabetes Association. 11. Microvascular Complications and Foot Care: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S135-S151. doi: 10.2337/dc20-S011. PMID 31862754
- [Result] American Diabetes Association. 6. Glycemic Targets: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S66-S76. doi: 10.2337/dc20-S006. PMID 31862749
- [Result] Phelan H, Lange K, Cengiz E, Gallego P, Majaliwa E, Pelicand J, Smart C, Hofer SE. ISPAD Clinical Practice Consensus Guidelines 2018: Diabetes education in children and adolescents. Pediatr Diabetes. 2018 Oct;19 Suppl 27:75-83. doi: 10.1111/pedi.12762. No abstract available. PMID 30175451
- [Result] Viana LV, Gomes MB, Zajdenverg L, Pavin EJ, Azevedo MJ; Brazilian Type 1 Diabetes Study Group. Interventions to improve patients' compliance with therapies aimed at lowering glycated hemoglobin (HbA1c) in type 1 diabetes: systematic review and meta-analyses of randomized controlled clinical trials of psychological, telecare, and educational interventions. Trials. 2016 Feb 17;17:94. doi: 10.1186/s13063-016-1207-6. PMID 26888087
- [Result] Sun C, Malcolm JC, Wong B, Shorr R, Doyle MA. Improving Glycemic Control in Adults and Children With Type 1 Diabetes With the Use of Smartphone-Based Mobile Applications: A Systematic Review. Can J Diabetes. 2019 Feb;43(1):51-58.e3. doi: 10.1016/j.jcjd.2018.03.010. Epub 2018 Mar 27. PMID 30026048